CLINICAL TRIAL: NCT00807950
Title: Phase II Study of Simvastatin in Primary Breast Cancer; Test of Its Potential Selectivity on Basal Subtype Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Purpose: Treatment
Other Study IDs: BR04/18/08
Record Dates: First submitted 2008-12-11; First posted 2008-12-15 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
We hypothesize that Simvastatin administration would result in selective killing of the basal subtype of breast cancer, in particular, CD44+/CD24- breast cancer cells in primary tumor. We further hypothesize that tumor genomic changes would correlate with tumor response to Simvastatin. We are also looking to correlate Simvastatin biological effects with the expression pattern of initial status of primary tumor. In addition, we hypothesize that Simvastatin-induced tumor gene expression changes may correlate with tumor and plasma proteomics, peripheral blood mononuclear cell gene expression changes, and pharmacogenetics, and that these analyses may further refine the selection of patients most likely to benefit from Simvastatin.

DETAILED DESCRIPTION:
Primary Objectives

1. Evaluate the biological response (proliferation and apoptosis) of Simvastatin in primary breast cancer.

2. Evaluate the cell type specificity of Simvastatin effect on basal subtype breast cancer, especially cells with CD44+/CD24- immunophenotype in the primary tumor. Secondary objectives

1. To study cellular response to Simvastatin in transriptome.
2. To obtain gene expression signature that predict Simvastatin biological effects.
3. To identify genetic polymorphisms that may influence Simvastatin pharmacokinetics and/or biological effects on breast cancer.
4. To correlate tumor and plasma proteomics with tumor gene expression changes, and to identify tumor and/or serum protein markers that predict Simvastatin biological effects.
5. To correlate peripheral blood mononuclear cell gene expression changes with tumor gene expression changes, and to identify blood gene markers that may predict Simvastatin biological effects. VI. Abstract of Research Proposal In no more than 300 words, describe concisely the specific aims, hypotheses, methodology and approach of the application, indicating where appropriate the application's importance to science or medicine. The abstract must be self-contained so that it can serve as a succinct and accurate description of the application when separated from it. Please use lay terms. If this not possible, the technical and medical terms should be explained in simple language. We hypothesize that Simvastatin administration would result in selective killing of the basal subtype of breast cancer, in particular, CD44+/CD24- breast cancer cells in primary tumor. We further hypothesize that tumor genomic changes would correlate with tumor response to Simvastatin. We are also looking to correlate Simvastatin biological effects with the expression pattern of initial status of primary tumor. In addition, we hypothesize that Simvastatin-induced tumor gene expression changes may correlate with tumor and plasma proteomics, peripheral blood mononuclear cell gene expression changes, and pharmacogenetics, and that these analyses may further refine the selection of patients most likely to benefit from Simvastatin. This is a single-centre, open-label, phase II study of Simvastatin in resectable primary breast cancer.

A total of 100 patients with measurable, resectable, primary breast tumor will be enrolled to receive 10-21 days of Simvastatin at a dose of 20 mg daily before definitive breast cancer surgery. Pre-treatment tumor biopsy will be obtained from each subject before starting Simvastatin. Subjects will take Simvastatin at a dose of 20 mg daily for 10-21 days, prior to definitive breast cancer surgery. The post-treatment tumor biopsy will be obtained at surgery. At each tumor biopsy, 3-4 tumor samples will be obtained through the same needle track. One tumor core at each time point will be fixed in formalin for histological examination and immunohistochemical studies. The remaining tumor cores will be stored in liquid nitrogen for subsequent RNA and protein extraction for gene expression and proteomics studies. Blood samples will be obtained before and after 10-21 days of Simvastatin treatment for Simvastatin pharmacokinetic analysis, plasma proteomics and peripheral mononuclear cell gene expression analysis. 10 ml blood will be taken from each participant for genotyping studies.

ELIGIBILITY:
Inclusion Criteria:

* Female, age >= 18 years. Page 14 of 28
* Histologic or cytologic diagnosis of breast carcinoma.
* Clinical T1-3 breast cancer with measurable primary breast tumor which is amenable to free-hand core biopsy
* Patients scheduled for definitive surgery
* Patients must not have received prior or scheduled to receive chemotherapy, hormonal therapy, radiotherapy, targeted therapy, or immunotherapy for the treatment of breast cancer.
* Karnofsky performance status of 70 or higher.
* Normal creatinine kinase
* Adequate organ function including the following:
* Bone marrow:
* Absolute neutrophil (segmented and bands) count (ANC) >= 1.5 x 109/L Platelets >= 100 x 109/L
* Hepatic:
* Bilirubin within normal range
* ALT or AST <1.5 x upper limit normal
* Renal:
* creatinine <= 1.5 x upper limit normal
* Signed informed consent from patient or legal representative.
* Patients with reproductive potential must use an approved contraceptive method if appropriate (eg, intrauterine device, birth control pills, or barrier device) during and for three months after the study. Females with childbearing potential must have a negative pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

* Current treatment with HMG-CoA reductase inhibitors or other lipid lowering drugs
* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Known hypersensitivity to Simvastatin
* Active liver disease or unexplained persistent elevations of serum transminases
* Pregnancy.
* Breast feeding
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2008-03; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Kumar AS, Benz CC, Shim V, Minami CA, Moore DH, Esserman LJ. Estrogen receptor-negative breast cancer is less likely to arise among lipophilic statin users. Cancer Epidemiol Biomarkers Prev. 2008 May;17(5):1028-33. doi: 10.1158/1055-9965.EPI-07-0726. Epub 2008 May 7. PMID 18463402
- [Background] Campbell MJ, Esserman LJ, Zhou Y, Shoemaker M, Lobo M, Borman E, Baehner F, Kumar AS, Adduci K, Marx C, Petricoin EF, Liotta LA, Winters M, Benz S, Benz CC. Breast cancer growth prevention by statins. Cancer Res. 2006 Sep 1;66(17):8707-14. doi: 10.1158/0008-5472.CAN-05-4061. PMID 16951186
- [Derived] Wang T, Seah S, Loh X, Chan CW, Hartman M, Goh BC, Lee SC. Simvastatin-induced breast cancer cell death and deactivation of PI3K/Akt and MAPK/ERK signalling are reversed by metabolic products of the mevalonate pathway. Oncotarget. 2016 Jan 19;7(3):2532-44. doi: 10.18632/oncotarget.6304. PMID 26565813